CLINICAL TRIAL: NCT06617715
Title: A Phase Ⅲ Clinical Study to Evaluate the Safety and Immunogenicity of 13-Valent Pneumococcal Conjugate Vaccine (PCV13) in Healthy Infants
Brief Title: Clinical Trial of 13-Valent Pneumococcal Conjugate Vaccine
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-PCV-3001
Record Dates: First submitted 2024-09-26; First posted 2024-09-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pneumococcal Infectious Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Sinovac PCV13 (Experimental): Participants aged 6 weeks-5 years will receive 4 doses of Sinovac PCV13 according to different immunization schedules.
  Interventions: Biological: Sinovac PCV13
- Active Comparator: Prevnar® (Active Comparator): Participants aged 6 weeks-5 years will receive 4 doses of Prevnar 13® according to different immunization schedules.
  Interventions: Biological: Prevnar®

INTERVENTIONS:
Biological: Sinovac PCV13 — One dose of Sinovac PCV13 (0.5 mL) is administered intramuscularly.
  Arms: Experimental: Sinovac PCV13
Biological: Prevnar® — One dose of Prevnar® (0.5 mL) is administered intramuscularly.
  Arms: Active Comparator: Prevnar®

SUMMARY:
A Phase Ⅲ clinical trial of 13-valent pneumococcal conjugate vaccine (PCV13) developed by Sinovac Life Science Co., Ltd will be conducted in pediatric population aged 2 months (minimum 6 weeks)-5 years (before 6th birthday). The objective of the study is to evaluate the immunogenicity and safety of Sinovac PCV13.

DETAILED DESCRIPTION:
A phase Ⅲ clinical trial of the study of 13-valent Pneumococcal Polysaccharide Conjugate Vaccine (PCV13) developed by Sinovac Life Science Co., Ltd (Sinovac) will be conducted in Chinese pediatric population aged 2 months (minimum 6 weeks)-5 years (before the 6th birthday). The trial is a randomized, double-blind, active controlled study. The objective of this study is to evaluate the immunogenicity and safety of PCV13 manufactured by Sinovac Life Science Co., Ltd. The active control vaccine is Prevenar13®. A total of at least 3080 participants aged 6 weeks to 5 years will be enrolled. Participants will be randomized in 1:1 ratio to the test group or control group.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants or children who are aged 2 months (at least 6 weeks), 7-11 months, 12-23 months and 2-5 years (before the 6th birthday);
2. Participants' guardians provide legal identity document and participants' vaccination record;
3. Participants' guardians understand and voluntarily sign the informed consent form;
4. Participants' guardians can follow all study procedures and stay in contact during the study.

Exclusion Criteria:

1. Received any pneumococcal vaccine prior to enrollment;
2. History of bacterial pneumonia or invasive pneumococcal diseases (IPDs) caused by Streptococcus pneumoniae, as confirmed by laboratory tests;
3. History of allergy or adverse reactions to the vaccine or vaccine components, or history of allergy, such as urticaria, dyspnea, angioedema and abdominal pain;
4. History of dystocia, asphyxia rescue and nervous system damage at birth for infants under 2 years of age;
5. Congenital malformations or developmental disorders, genetic defects, severe malnutrition, history of asthma;
6. Autoimmune diseases (such as systemic lupus erythematosus), immunodeficiency diseases or immunosuppressive diseases (such as AIDS, organ transplantation);
7. Severe cardiovascular diseases, diabetes, liver diseases, kidney diseases, malignant tumours.
8. Have/have suffered from a serious neurological disorder (epilepsy or convulsions) or mental illness or have a family history of such diseases.
9. History of thyroidectomy, asplenia, functional asplenia; asplenia or splenectomy caused by any reasons;
10. Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets level), history of obvious bleeding, hematoma or bruising after intramuscular injection or venipuncture.
11. Consecutively received ≥14 days of corticosteroid, any other immunosuppressive therapy (excluding corticosteroid spray therapy for allergic rhinitis and surface corticosteroid therapy for acute non-concurrent dermatitis), or cytotoxic therapy prior to enrollment for infants aged 6 weeks to 2 months or within 6 months prior to enrollment for children aged 7 months to 5 years.
12. Received blood products prior to enrollment for children aged 2 months or within 3 months prior to enrollment for children aged 7 months to 5 years. Receipt of Hepatitis B immunoglobulin one month prior to enrollment is an exception.
13. Received other investigational drugs within 60 days prior to enrollment, or plan to receive such drugs during the study;
14. Received live attenuated vaccine within 14 days prior to enrollment;
15. Received subunit or inactivated or other vaccine within 7 days prior to enrollment;
16. Acute diseases or acute onset of chronic diseases within 7 days prior to enrollment;
17. Had fever (axillary temperature≥ 37.3 Degree Celsius) before vaccination;
18. In the investigator's judgment, the participant has any other factors that make him or her unfit to participate in the clinical trial.

Ages: 6 Weeks to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3080 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-05-12 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of pneumococcal serotype-specific IgG antibody concentration ≥0.35 μg/ml (seropositive rate) | 30 days after primary vaccination
  Proportion of serotype-specific IgG concentration ≥0.35 μg/ml
Pneumococcal serotype-specific IgG antibody geometric mean concentration (GMC) | 30 days after primary vaccination
  IgG GMC

SECONDARY OUTCOMES:
Proportion of pneumococcal serotype-specific IgG antibody concentration ≥0.35 μg/ml (seropositive rate) | 30 days after booster vaccination
  Proportion of serotype-specific IgG concentration ≥0.35 μg/ml
Pneumococcal serotype-specific IgG antibody geometric mean concentration (GMC) | 30 days after booster vaccination
  IgG GMC
Proportion of pneumococcal serotype-specific OPA antibody GMT≥1:8 | 30 days after primary vaccination
  Proportion of participants with pneumococcal serotype-specific OPA antibody titers ≥ 1:8
Pneumococcal serotype-specific OPA antibody geometric mean titer (GMT) | 30 days after primary vaccination
  Pneumococcal serotype-specific OPA antibody GMT
Proportion of participants with a pneumococcal serotype-specific IgG concentration ≥ 1.0 μg/mL | 30 days after primary vaccination
  Proportion of participants with a pneumococcal serotype-specific IgG concentration ≥ 1.0 μg/mL
Pneumococcal serotype-specific IgG antibody geometric mean increase (GMI) | 30 days after primary vaccination
  Pneumococcal serotype-specific IgG GMI
Pneumococcal serotype-specific OPA antibody geometric mean increase(GMI) | 30 days after primary vaccination
  Pneumococcal serotype-specific OPA antibody GMI
Proportion of participants with a pneumococcal serotype-specific IgG concentration ≥ 1.0 μg/mL | 30 days after booster vaccination
  Proportion of participants with a pneumococcal serotype-specific IgG concentration ≥ 1.0 μg/mL
Pneumococcal serotype-specific IgG antibody geometric mean increase (GMI) | 30 days after booster vaccination
  Pneumococcal serotype-specific IgG GMI
Proportion of participants with pneumococcal serotype-specific OPA titers ≥ 1:8 (seropositive rate) | 30 days after booster vaccination
  Proportion of participants with pneumococcal serotype-specific OPA titers ≥ 1:8 (seropositive rate)
Pneumococcal serotype-specific OPA antibody geometric mean titer (GMT) | 30 days after booster vaccination
  Pneumococcal serotype-specific OPA antibody GMT
Pneumococcal serotype-specific OPA antibody geometric mean increase(GMI) | 30 days after booster vaccination
  Pneumococcal serotype-specific OPA antibody GMI
Safety of Sinovac PCV13 | 0-30 days within each dose
  Incidence of adverse reactions
Safety of Sinovac PCV13 | 6 months within final dose
  Incidence of serious adverse events

OTHER OUTCOMES:
Proportion of participants with a pneumococcal serotype-specific IgG concentration ≥ 0.35 μg/mL (seropositive rate) | 1,2,3 years after final dose
  Proportion of participants with a pneumococcal serotype-specific IgG concentration ≥ 0.35 μg/mL (seropositive rate)
Proportion of participants with a pneumococcal serotype-specific IgG concentration ≥ 1.0 μg/mL | 1,2,3 years after final dose
  Proportion of participants with a pneumococcal serotype-specific IgG concentration ≥ 1.0 μg/mL
Pneumococcal serotype-specific IgG geometric mean concentration (GMC) | 1,2,3 years after final dose
  Pneumococcal serotype-specific IgG geometric mean concentration (GMC)
Proportion of participants aged 2-5 years with pneumococcal serotype-specific OPA titers ≥ 1:8 (seropositive rate) | 1,2,3 years after vaccination
  Proportion of participants aged 2-5 years with pneumococcal serotype-specific OPA titers ≥ 1:8
Pneumococcal serotype-specific OPA antibody geometric mean titer (GMT) in participants aged 2-5 years | 1,2,3 years after vaccination
  Pneumococcal serotype-specific OPA antibody GMT in participants aged 2-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Wang, Principal Investigator — Henan Provincial Center for Disease Control and Prevention
Locations (1):
- Henan Provincial Center for Disease Control and Prevention, Zhengzhou, Henan, China